CLINICAL TRIAL: NCT00268099
Title: Optimal Timing for Repair of Right-to-Left Shunt Lesions
Status: Terminated | Type: Observational
Why Stopped: study not started
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-121
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-06

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; repair of right to left shunt lesions; Tetralogy of Fallot defects
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of this study is to determine the optimal timing for repair of right-to-left shunt lesions such as Tetralogy of Fallot defects.

The secondary aim being define the criteria for failing medical therapy.

DETAILED DESCRIPTION:
In the past, children with right-to-left shunt lesions such as Tetralogy of Fallot defects were palliated with a systemic to pulmonary artery shunt. This prevented cyanosis while the child grew to a size where complete repair could be undertaken. With the improvements in surgical technique and critical care, there is a push to do a primary complete repair for these defects at younger and younger ages. These operations should be delayed as long as possible to allow for growth but not so long that there is unnecessary cyanosis and hypoxemia.

Study Design and Methodology:

Retrospective chart review - approximately 75 patients

Preoperative data:

Diagnosis

Operative data:

Age and weight at surgery Type of surgical procedure Whether pulmonary valve is spared

Postoperative data:

Length of time on ventilator Length of time on inotropes Length of ICU stay Length of hospital stay Complications

ELIGIBILITY:
Inclusion Criteria:

* patients in the congenital surgery database who have undergone repair of a Tetralogy of Fallot defect

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients in the congenital surgery database who have undergone repair of a Tetralogy of Fallot defect
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2005-05; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States